CLINICAL TRIAL: NCT06477575
Title: Effectiveness of Technology-based Interventions for the Improvement of Cognitive Processes in Children and Adolescents With ADHD.
Brief Title: Effectiveness of Technology-based Interventions for the Improvement of Cognitive Processes in ADHD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Clinical Proffesor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210624
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: ADHD, Deficits in Motor Control and Perception
Keywords: ADHD; cognitive rehabilitation; new technologies
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neurocognitive therapy based on new technologies (Experimental)
  Interventions: Device: neurocognitive therapy based on new technologies
- conventional neurocognitive therapy (Active Comparator)
  Interventions: Other: conventional neurocognitive therapy

INTERVENTIONS:
Device: neurocognitive therapy based on new technologies — The cognitive neurorehabilitation program is based on gaming through the use of the Nintendo Switch device. The following games have been chosen: Pufferfish, Hex Egg, Mystic Totem, Thor's Thunder, since they are games that work on selective attention, concentration and processing speed, which are the variables to be studied in this project.
  Hardware: Nintendo Switch Software: 60 in 1 game Games: Pufferfish, Hex Egg, Mystic Totem, Thor's Thunder. Therapy time: 30 minutes effective. Number of Sessions: 2 per week / Number of weeks: 8 Total number of intervention sessions: 16 sessions Place: Thercli Center (Don Benito).
  Arms: neurocognitive therapy based on new technologies
Other: conventional neurocognitive therapy — The cognitive neurorehabilitation program for group active comparator is based on playing more conventional board games that work on selective attention, concentration and processing speed, which are the variables to be studied in this project.
  Traditional games and token book. Games: Dobble, Lynx, Crazy cups, Jungle speed, animalea, ghost. Card: Stimulate and learn level 3 and 4. Therapy time: 30 minutes effective. No. of sessions: 2 per week / No. of weeks: 8 Total number of intervention sessions: 16 sessions Place: Thercli Center (Don Benito).
  Arms: conventional neurocognitive therapy

SUMMARY:
To scientifically demonstrate the improvements in cognitive functions and core symptoms of children and adolescents diagnosed with ADHD through the implementation of a cognitive rehabilitation program based on the use of the most relevant technologies found in the systematic review carried out during the first phase.

Two intervention groups will be randomly assigned for the study:

G1: composed of 20 patients who will receive neurocognitive therapy based on new technologies. This will be the experimental group.

G2: composed of 20 patients who will receive conventional neurocognitive therapy for ADHD treatment. This group will be the control group

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents diagnosed with ADHD
* Age: 6-17 years old

Exclusion Criteria:

* Children and adolescents diagnosed with ADHD + ADD.
* Age: under 6 years old or over 17 years old.
* Other psychopharmacological treatments not specific for ADHD.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
WisC-V (Wechsler intelligence scale for children) | 8 weeks
  provides primary intelligence index scores that reflect intellectual functioning in different cognitive areas: verbal comprehension, visuospatial, fluid reasoning, working memory and processing speed.
STROOP (Colors and Words Test) | 8 weeks
  reference test for the detection of neuropsychological problems and brain damage. It allows to evaluate the phenomenon of interference, intimately linked to inhibitory control processes.
CARAS-R(Difference perception test) | 8 weeks
  evaluates the ability to quickly and correctly perceive similarities and differences in partially ordered patterns of stimulation. It measures perceptual and attentional skills by means of 60 graphic items consisting of schematic drawings of faces with elementary strokes.

CONTACTS AND LOCATIONS:
Locations (1):
- Berta Caro Puértolas, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No